CLINICAL TRIAL: NCT03960619
Title: In Person and Mobile Health Coping Skills Training for Improving Symptom Management and Daily Steps in Hematopoietic Stem Cell Transplant Patients
Acronym: CST Step Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00100451
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hematopoietic Neoplasms (Leukemia, Lymphoma, Multiple Myeloma)
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- in-person & mHealth coping skills training (Experimental): hybrid in-person and mHealth coping skills training and activity coaching intervention is to reduce physical disability and decrease pain, fatigue and stress while enhancing patients' abilities to cope with symptoms that interfere with activity.
  Interventions: Behavioral: coping skills training

INTERVENTIONS:
Behavioral: coping skills training — We aim to test a combined coping skills training and activity coaching protocol that: first, is feasible and acceptable, and second, improves physical disability, as well as pain, fatigue, distress, and physical activity in HCT patients. We propose a novel intervention protocol that uses a hybrid in-person and mHealth intervention delivery model.

SUMMARY:
The purpose of the study is to assess the feasibility, acceptability, and efficacy of a novel mHealth behavioral intervention to enable HCT patients to effectively cope with symptoms to improve their ability to engage in physical activity that can improve physical disability. Our interdisciplinary team (psychiatry, hematology/oncology, occupational therapy) proposes a single arm pilot trial (N=20) to test a hybrid in-person and mHealth (video-conferencing, symptoms/activity monitoring, personalized feedback via text) HCT Coping Skills Training for Symptom Management and Daily Steps (CST Step-Up) intervention. CST Step-Up will provide patients with coping skills training and activity coaching sessions to enhance their ability to cope with symptoms that interfere with activity.

DETAILED DESCRIPTION:
Our group developed a mHealthpain coping skills training program for HCT patients and found in a small pilot trial (R21) that improved pain coping led to increased daily activity and reduced physical disability. However, fatigue and distress were also barriers to physical activity.

We propose to assess the feasibility, acceptability, and outcome patterns suggesting efficacy of a novel mHealth behavioral intervention to enable HCT patients to effectively cope with symptoms to improve their ability to engage in physical activity that can improve physical disability.Our interdisciplinary team (psychiatry, hematology/oncology, occupational therapy) is conducting a single arm pilot trial (N=20) to test a hybrid in-person and mHealth (video-conferencing, symptoms/activity monitoring, personalized feedback via text) HCT Coping Skills Training for Symptom Management and Daily Steps (CST Step-Up) intervention. CST Step-Up will provide patients with coping skills training and activity coaching sessions to enhance their ability to cope with symptoms that interfere with activity.

Aim 1:Use a single arm pilot trial (N=20) to examine the feasibility and acceptability of the CST Step-Up protocol. Feasibility will be assessed via (a) study accrual, (b) adherence to the study protocol (intervention and assessments), and (c) retention (% completing the study).

H1:Feasibility will be determined by meeting targeted study accrual (20 patients 15 months), >80% adherence to the protocol, and <20% attrition. Acceptability will be demonstrated by 80% of participants reporting satisfaction with the intervention.

Aim 2:Examine outcome patterns suggesting the efficacy of the CST Step-Up protocol for improving physical disability and other important outcomes.

H2:Pre-and post-intervention differences will be examined with simple t-tests to evaluate patterns suggesting intervention efficacy on measures of physical disability (self-report, 6-min walk test), pain, fatigue, distress, physical activity (daily steps), and self-efficacy for symptom management.

Confirmed hypotheses would provide the first demonstration of the feasibility, acceptability, and positive impact of a hybrid in-person and mHealth coping skills training and activity coaching intervention that reduces physical disability by concurrently and synergistically decreasing symptom burden and increasing physical activity. This project has the potential to lead to future research (e.g., R01) that can redesign existing modes of behavioral intervention delivery, improve continuity and coordination of care, and ultimately enhance patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* undergone hematopoietic stem cell transplant (HCT) due to an oncological disease (e.g., leukemia, lymphoma, multiple myeloma)
* being at least 18years old and
* life expectancy at least 12 months.

Exclusion Criteria:

* cognitive impairment (e.g., dementia) recorded in the chart or suspected by healthcare provider,
* presence of a severe psychiatric condition (i.e., psychotic disorder or episode) or a psychiatric condition (e.g., suicidal intent) that would contraindicate safe participation in the study as indicated by the medical chart, treating oncologist, or interactions with the medical/study staff, and
* inability to converse in English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Accrual as measured by number of participants recruited | 15 months
  Accrual will be indicated by meeting the recruitment goal
Adherence as measured by completing all intervention sessions | 15 months
  Adherence will be indicated by the proportion successfully completing intervention sessions
Attrition as measured by 80% participants completing the study. | 15 months
  Attrition will be indicated by 80% of consented participants completing the study protocol.
Acceptability as measured by 80% participants reporting satisfaction with CST program | 15 months
  Acceptability will be indicated by 80% of patients reporting satisfaction with CST Step-Up on the CSQ.

SECONDARY OUTCOMES:
Change in Physical Disability | assessments at baseline (pre - treatment) and post-intervention at 3-months..
  Functional Assessment of Cancer Therapy 7-item physical well-being scale will be used to assess physical disability.
Change in Fatigue | assessments at baseline (pre-treatment) and post-intervention at 3-months.
  Fatigue will be measured with the PROMIS Adult Fatigue Short Form.
Change in Psychological Distress | assessments at baseline (pre-treatment) and post-intervention at 3-months.
  Psychological Distress will be measured with the Brief Symptom Inventory
Change in Self-Efficacy for Symptom Management: PROMIS Self-Efficacy for Managing Symptoms Short Form | assessments at baseline (pre-treatment) and post-intervention at 3-months.
  Self-Efficacy for Symptom Management will be measured with the PROMIS Self-Efficacy for Managing Symptoms Short Form
Symptom Monitoring | post-intervention at 3-months.
  Symptom Monitoring will involve participants using the study phone to provide (text) daily average ratings of Pain, fatigue, and distress on a 0=none to 10=worst imaginable scale. Symptom data will inform personalized feedback via text from the therapist to the CST Step-Up participant.
Physical Activity | post-intervention at 3-months.
  Physical Activity will be measured by asking participants to monitor daily activity as assessed by step count with a wireless activity tracker (e.g., Fitbit) that syncs with assigned study phone.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara J Somers, PhD, Principal Investigator — Duke University
Locations (1):
- Duke university health system, Durham, North Carolina, United States